CLINICAL TRIAL: NCT03730441
Title: Correlation Between ADR of Screening and All Colonoscopies
Status: Completed | Type: Observational
Sponsor: Hospital Frydek-Mistek (Other)
Responsible Party: Principal Investigator, Ivana Mikoviny Kajzrlikova, MD, PhD, MD, Hospital Frydek-Mistek
Other Study IDs: ADR
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Colon Neoplasm
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Colonoscopy — Endoscopic examination of large bowel

SUMMARY:
The aim of the study is to compare ADR for colonoscopies from various indications and to find correlations between ADR of screening and all examinations.

DETAILED DESCRIPTION:
ADR (adenoma detection rate) is generally accepted quality indicator and it is calculated from screening colonoscopies in patients over 50 years of age. For possible gaming with ADR for screening colonoscopies, monitoring of ADR for all colonoscopies is discussed nowadays.The aim of the study is to compare ADR for colonoscopies from various indications and to find correlations between ADR of screening and all examinations.

We want to retrospectively assess the quality indicators of all colonoscopies performed from January 2013 to December 2017. We want to calculate ADR for all colonoscopies in patients over 50 years of age excluding therapeutic, IBD, management of complications and sigmoidoscopies (screening, surveillance, diagnostic) and separately only for screening colonoscopies. Correlation analysis will be performed using Pearson´s correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* people over 50 years of age coming for colonoscopic examination (screening, surveillance, diagnostic)

Exclusion Criteria:

* age under 50 years
* indication for colonoscopy: therapeutic, IBD, management of complications and sigmoidoscopies

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people over 50 years of age coming for colonoscopic examination
Sampling Method: Probability Sample
Enrollment: 6925 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
correlation between ADR of screening and all colonoscopies (screening, surveillance, diagnostic) | january 2013 - december 2017
  Pearson´s correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Mikoviny Kajzrlikova, Principal Investigator — Doctor
Locations (1):
- Hospital Frydek-Mistek, Frýdek-Místek, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
ADRs of all endoscopists in our unit for both all and screening colonoscopies

REFERENCES:
- [Derived] Mikoviny Kajzrlikova I, Vitek P, Chalupa J, Kuchar J, Platos J, Reha P, Klvana P. Correlation between ADR of screening and all colonoscopies. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2021 Nov;165(4):386-389. doi: 10.5507/bp.2020.059. Epub 2020 Dec 16. PMID 33325459